CLINICAL TRIAL: NCT02941614
Title: Implementing Systematic Distress Screening in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: California Breast Cancer Research Program (Other)
Responsible Party: Sponsor
Other Study IDs: KPSC IRB 11103
Record Dates: First submitted 2016-10-17; First posted 2016-10-21 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention: Newly diagnosed breast cancer patients will be offered a brief distress screening questionnaire, the Patient Health Questionnaire (PHQ), around the time of their breast cancer diagnosis and again at subsequent transitions in care as appropriate (e.g., the initiation of chemotherapy).
  Interventions: Behavioral: Distress screening
- Control: Newly diagnosed breast cancer patients will experience usual care.

INTERVENTIONS:
Behavioral: Distress screening — A brief depression and anxiety screening instrument, the Patient Health Questionnaire-9 (PHQ-9), will be administered to newly diagnosed breast cancer patients in the Distress Screening arm.
  Groups: Intervention

SUMMARY:
Many breast cancer patients experience psychological distress during their cancer care journey. There are effective treatments for breast cancer patients experiencing distress, such as individual or group therapy, health education, and medication. Unfortunately, clinicians may not be aware of the symptoms of distress in their breast cancer patients, and some breast cancer patients who could benefit from referral to behavioral health specialists are overlooked. New guidelines recommend that all cancer patients be regularly screened for distress. However, there are unanswered questions about the impact of distress screening conducted on a large scale. Few studies have evaluated the impact of distress screening on important outcomes in breast cancer patients, such as patient experience and use of health care services, as compared to the usual care offered by the health care organization. In addition, oncology clinicians may be uncertain about the benefits of large-scale distress screening, and pilot screening programs have not been uniformly successful particularly in the community oncology setting.

The overarching goals of this study are to assess the effectiveness of implementing a guideline-recommended distress screening program for newly diagnosed breast cancer patients on improving identification and referral to treatment for highly distressed breast cancer patients, to assess patient-reported outcomes, health services utilization, and implementation outcomes of the program. This study will address two main research questions: 1) Evaluate the effectiveness of a guideline-recommended distress screening program for breast cancer patients in improving identification of distressed patients, initiation and completion of referrals to behavioral health, and patient-reported and utilization outcomes as compared to usual care; 2) Identify the barriers, facilitators, and other implementation-related outcomes related to distress screening in the community oncology setting.

Please note: This study did not require a DSMB, as it falls under the exception for low-risk behavioral studies.

DETAILED DESCRIPTION:
Background and Study Aims:

Breast cancer patients are at risk for physical and psychosocial harms. Among the most highly prevalent psychosocial issues in breast cancer patients is psychological distress. Distress is defined and assessed as psychiatric morbidity or prevalence of psychiatric disorders, particularly anxiety and depression. It is estimated that 40-50% of women diagnosed with early stage breast cancer will experience distress in the year following diagnosis. There is a rich literature on the persistent negative effects of distress in breast cancer patients, including associations with decreased physical and social functioning, increased symptom burden, higher utilization of inpatient and emergency services, and poor quality of life. Psychological distress can also adversely affect individual work productivity, and contributes to the rising costs of cancer care.

Recent guidelines from the American Society of Clinical Oncology (ASCO) and others recommend routine distress screening for breast cancer patients, recognizing the availability of effective treatments for psychological distress. Unfortunately distress remains under-detected and undertreated in breast cancer patients and rates of adherence to ASCO and other guidelines is very low. Low rates of screening might be explained in part by limited evidence of effectiveness: while efficacy of distress screening has been demonstrated in small-scale trials at academic centers, typically showing increases in number of referrals to psychosocial services, evidence supporting the effectiveness of large scale distress screening programs under routine practice conditions is limited. It is currently unknown if distress screening of breast cancer patients will improve identification of distressed patients or referrals to behavioral health services in non-academic settings. In addition, extant efficacy studies generally fail to measure key impacts and outcomes desired from distress screening, such as patient-reported outcomes (e.g., distress management, satisfaction) and changes in health care utilization (e.g., changes in emergency department use). Implementation-related factors and outcomes have also been largely overlooked in prior research (e.g., clinician acceptability, fidelity of delivery), leaving serious gaps in the understanding of barriers to adoption of distress screening programs and gaps in the knowledge needed to facilitate large-scale, routine implementation of screening.

The overarching goal of this study is to implement and evaluate a guideline-based distress screening program for newly diagnosed breast cancer patients, measuring its effectiveness and impacts on key outcomes and examining barriers and facilitators to routine adoption. There is a critical need for translational research to assess the effectiveness of distress screening programs in improving (a) identification of distress, (b) referral for services, (c) outcomes for breast cancer patients in real-world oncology settings, and in understanding implementation barriers and facilitators. Without evidence of effectiveness, it is unlikely that clinical and operational health system leaders will invest in distress screening programs, potentially leading to serious adverse consequences. This proposed translational research is crucial in order to bridge the gap between academic studies and non-academic, community oncology practice, where the majority of breast cancer patients are treated. In addition, gaining insight and understanding into barriers and facilitators to implementation of distress screening programs is critically important. The objectives are to assess the effectiveness of the recommended screening program from the joint task force of the American Psychosocial Oncology Society, Association of Oncology Social Work, and Oncology Nursing Society on improving identification and referral to treatment for highly distressed breast cancer patients within an integrated health care system, and to assess patient-reported outcomes, health services utilization, and implementation outcomes of the program.

Specific Aims:

Aim 1: Evaluate the effectiveness of a guideline-recommended distress screening program for breast cancer patients in improving identification of distressed patients, initiation and completion of referrals to behavioral health, and patient-reported and utilization outcomes as compared to usual care within Kaiser Permanente Southern California (KPSC), using a pragmatic cluster randomized control trial design at six medical centers.

Aim 2: Identify patient-, clinician-, and system-level barriers and facilitators to implementation of the program, and assess stakeholder-perceived acceptability, fidelity, and achievements of the program.

Study Methods The setting for this research is Kaiser Permanente Southern California, a large, integrated health care system with 14 medical centers serving a highly diverse population of over 4 million members. The investigators will use a novel hybrid effectiveness-implementation study design that allows for dual study of the clinical effectiveness and implementation-related factors to address the need for evidence in both areas. This study will employ mixed methods, collecting both qualitative and quantitative data as appropriate to address the study aims. To evaluate effectiveness, this study will use a cluster randomized control trial (RCT) design, clustered at the medical center level, and will implement the program at the intervention sites and offering screening to all newly diagnosed breast cancer patients. To evaluate the effectiveness of the program, the investigators will collect structured data from the KPSC electronic record (referral initiation/completion, use of health services) and patient-reported data (functioning, symptom management). Existing work from a pilot primary care-based distress screening program will be leveraged for this research, demonstrating the feasibility of this study. Implementation outcomes will be assessed with qualitative and survey data.

Knowledge gained from this research will be used to inform the continued development and implementation of systematic distress screening programs for breast cancer patients, and will enrich the evidence base by providing critical information on relevant patient- and system-level outcomes. These results will have an impact on the quality of life and quality of care for these patients, and will directly influence distress screening program adoption, scale-up, and spread, making this work highly relevant to breast cancer patients throughout California and across the nation.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with initial breast cancer, any stage, any histology type
* Kaiser Permanente member for at least 100 days during study period

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 1436 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin E Hahn, PhD, Principal Investigator — Kaiser Permanente
Locations (6):
- United States (6):
  - Anaheim Medical Center, Anaheim, California
  - Baldwin Park Medical Center, Baldwin Park, California
  - South Bay - Harbor City Medical Center, Harbor City, California
  - Los Angeles Medical Center, Los Angeles, California
  - West Los Angeles Medical Center, Los Angeles, California
  - Woodland Hills Medical Center, Woodland Hills, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hahn EE, Munoz-Plaza CE, Lyons LJ, Lee JS, Pounds D, La Cava S, Brasfield FM, Durna LN, Kwan KW, Beard DB, Ferreira A, Gould MK. Barriers and facilitators to implementation and sustainment of guideline-recommended depression screening for patients with breast cancer in medical oncology: a qualitative study. Support Care Cancer. 2023 Jul 12;31(8):461. doi: 10.1007/s00520-023-07922-0. PMID 37436477
- [Derived] Hahn EE, Munoz-Plaza CE, Pounds D, Lyons LJ, Lee JS, Shen E, Hong BD, La Cava S, Brasfield FM, Durna LN, Kwan KW, Beard DB, Ferreira A, Padmanabhan A, Gould MK. Effect of a Community-Based Medical Oncology Depression Screening Program on Behavioral Health Referrals Among Patients With Breast Cancer: A Randomized Clinical Trial. JAMA. 2022 Jan 4;327(1):41-49. doi: 10.1001/jama.2021.22596. PMID 34982119

RESULTS

PARTICIPANT FLOW:
Groups:
- Distress Screening: Newly diagnosed breast cancer patients will be offered a brief distress screening questionnaire, the Patient Health Questionnaire (PHQ), around the time of their breast cancer diagnosis and again at subsequent transitions in care as appropriate (e.g., the initiation of chemotherapy).
  Distress screening: A brief depression and anxiety screening instrument, the Patient Health Questionnaire (PHQ-9) will be administered to newly diagnosed breast cancer patients in the Distress Screening arm.
- No Screening: Newly diagnosed breast cancer patients will experience usual care, which may include PHQ-9 screening.
Period: Overall Study
Arm/Group | Distress Screening | No Screening
Started | 744 | 692
Completed | 603 | 446
Not Completed | 141 | 246

BASELINE CHARACTERISTICS:
Groups:
- Distress Screening: Newly diagnosed breast cancer patients will be offered a brief distress screening questionnaire, the Patient Health Questionnaire (PHQ), around the time of their breast cancer diagnosis and again at subsequent transitions in care as appropriate (e.g., the initiation of chemotherapy).
  Distress screening: A brief depression and anxiety screening instrument, the Patient Health Questionnaire (PHQ), will be administered to newly diagnosed breast cancer patients in the Distress Screening arm. The PHQ starts with a 2-item screen, and branches to the full screening instrument as needed.
- No Screening: Newly diagnosed breast cancer patients will experience usual care.
- Total: Total of all reporting groups
Arm/Group | Distress Screening | No Screening | Total
Number analyzed (Participants) | 744 | 692 | 1436
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 425 | 381 | 806
  >=65 years | 319 | 311 | 630
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.35) | 62 (13.34) | 61.5 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 740 | 689 | 1429
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 204 | 172 | 376
  Not Hispanic or Latino | 483 | 476 | 959
  Unknown or Not Reported | 57 | 44 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 7 | 12
  Asian | 151 | 113 | 264
  Native Hawaiian or Other Pacific Islander | 6 | 7 | 13
  Black or African American | 106 | 143 | 249
  White | 401 | 370 | 771
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 73 | 50 | 123
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 744 | 692 | 1436
Charlson Comorbidity Score [Mean (Standard Deviation); unit: units on a scale] — The score included diagnoses from 1 year prior to the index visit and excluded codes for breast cancer. The index quantifies an individual's burden of disease corresponding 1-year mortality risk. 22 comorbid conditions are assessed, including heart disease, AIDS, cancer, etc. Each condition is assigned a score of 1, 2, 3, or 6 depending on the risk of dying associated with each one (1=lower risk; 6 = highest). Scores are summed to provide a total score to predict mortality.
  units on a scale | 2.2 (2.75) | 2.1 (2.62) | 2.2 (2.69)
Cancer Stage [Count of Participants; unit: Participants] — Cancer stage estimated from pathology, diagnosis codes, and visit notes. There are 5 stages of cancer assigned: stage 0 (carcinoma in situ), stage I, stage II, stage III and stage IV. Lower stages indicate that the disease is more localized, isolated or contained, whereas higher stages refer to cancers that have spread into other areas of the body. Stage 0 is considered the best outcome, with Stage IV representing the worst outcome.
  Participants
    Stage 0 | 32 | 27 | 59
    Stage I | 145 | 106 | 251
    Stage II | 236 | 234 | 470
    Stage III | 236 | 219 | 455
    Stage IV | 58 | 85 | 143
    Missing | 37 | 21 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Offered and Screened for Distress
Description: # of newly diagnosed breast cancer patients offered and screened with the Patient Health Questionnaire 9 at their initial consult
Time Frame: Patients assessed during initial consult - e.g. 1 day during 60 min consult
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Screening | No Screening
Number analyzed (Participants) | 744 | 692
Participants | 596 | 3

2. Primary Outcome: Number of Participants Offered an Appropriate Referral
Description: For patients who had screening done in Oncology, appropriate action for those with a medium/high PHQ-9 is a referral to social work, psychiatry, depression care management.
Time Frame: Patients assessed during initial consult - e.g. 1 day during 60 min consult
Population: Patients who completed PHQ-9 screening in Oncology with med/high score
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 63 | 1
Participants | 51 | 0

3. Secondary Outcome: Functional Assessment of Cancer Therapy, Breast Cancer (FACT-B)
Description: Self-reported for physical well-being; social family well-being; emotional well-being; functional well-being; and additional concerns over the past 7 days; scale: 0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much; responses indicate symptoms/concerns in the past 7 days. The higher the score, the better the outcome. To derive a FACT-B total score, score range 0-148. The subscales include: (1) Physical Well-Being, score range 0-28; (2) Social/Family Well-Being, score range 0-28; (3) Emotional Well-Being, score range 0-24; (4) Functional well-being, score range 0-28; (5) Breast Cancer Subscale, score range 0-40.
Time Frame: 12 months
Population: Patients who completed at least one survey item in Fact-B at the 3, 6 and/or 12 month survey. The number of participants analyzed for the total scores and sub-scale scores at 3-, 6- and 12 months varies, because not all patients responded to all surveys or answered all of the questions in a survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Distress Screening | No Screening
Number analyzed (Participants) | 224 | 238
units on a scale
  Fact-B 3-month Total Score: number analyzed (Participants) | 205 | 224
  Fact-B 3-month Total Score | 104.5 (22.1) | 104.6 (23.0)
  Fact-B 3-month Physical Well-Being Subscale: number analyzed (Participants) | 215 | 236
  Fact-B 3-month Physical Well-Being Subscale | 20.8 (6.2) | 20.5 (6.5)
  Fact-B 3 month Social/Family Well-Being Subscale: number analyzed (Participants) | 213 | 232
  Fact-B 3 month Social/Family Well-Being Subscale | 21.2 (6.2) | 21.4 (5.8)
  Fact-B 3 month Emotional Well-Being Subscale: number analyzed (Participants) | 220 | 232
  Fact-B 3 month Emotional Well-Being Subscale | 18.3 (4.3) | 18.3 (4.4)
  Fact-B 3-month Functional Well-Being Subscale: number analyzed (Participants) | 220 | 234
  Fact-B 3-month Functional Well-Being Subscale | 18.3 (6.7) | 18.1 (6.6)
  Fact-B 3-month Breast Cancer Subscale: number analyzed (Participants) | 215 | 232
  Fact-B 3-month Breast Cancer Subscale | 26.5 (6.8) | 26.4 (6.9)
  Fact-B 6 month Total Score: number analyzed (Participants) | 118 | 123
  Fact-B 6 month Total Score | 108.1 (22.3) | 105.3 (21.9)
  Fact-B 6 month Physical Well-Being Subscale: number analyzed (Participants) | 122 | 125
  Fact-B 6 month Physical Well-Being Subscale | 22.3 (5.9) | 21.9 (5.4)
  Fact-B 6 month Social/Family Well-Being Subscale: number analyzed (Participants) | 120 | 126
  Fact-B 6 month Social/Family Well-Being Subscale | 20.5 (6.2) | 21.3 (5.3)
  Fact-B 6 month Emotional Well-Being Subscale: number analyzed (Participants) | 120 | 126
  Fact-B 6 month Emotional Well-Being Subscale | 18.5 (4.3) | 18.0 (4.4)
  Fact-B 6 month Functional Well-Being Subscale: number analyzed (Participants) | 121 | 126
  Fact-B 6 month Functional Well-Being Subscale | 19.2 (6.2) | 18.5 (6.4)
  Fact-B 6 month Breast Cancer Subscale: number analyzed (Participants) | 120 | 125
  Fact-B 6 month Breast Cancer Subscale | 27.0 (6.9) | 25.8 (7.5)
  Fact-B 12 month Total Score: number analyzed (Participants) | 127 | 129
  Fact-B 12 month Total Score | 109.1 (22.9) | 108.3 (22.4)
  Fact-B 12 month Physical Well-Being Subscale: number analyzed (Participants) | 129 | 134
  Fact-B 12 month Physical Well-Being Subscale | 22.1 (5.6) | 22.3 (5.5)
  Fact-B 12 month Social/Family Well-Being Subscale: number analyzed (Participants) | 129 | 134
  Fact-B 12 month Social/Family Well-Being Subscale | 20.7 (6.1) | 20.9 (6.0)
  Fact-B 12 month Emotional Subscale: number analyzed (Participants) | 129 | 132
  Fact-B 12 month Emotional Subscale | 18.8 (3.9) | 18.6 (4.4)
  Fact-B 12 month Functional Well-Being: number analyzed (Participants) | 129 | 134
  Fact-B 12 month Functional Well-Being | 19.9 (6.3) | 19.9 (5.9)
  Fact-B 12 month Breast Cancer Subscale: number analyzed (Participants) | 130 | 132
  Fact-B 12 month Breast Cancer Subscale | 27.1 (6.9) | 26.9 (6.8)
Statistical Analysis 1: Comparison: Distress Screening vs No Screening; Data below is for FACT-B 3 month Total Score; Test type: Other — Conducted test of null hypothesis of no difference vs any, between intervention and control sites at three different time periods (6- vs. 3-months, 12- vs. 6-months, 12- vs. 3-months), as well as omnibus test of treatment-by-time interaction; p = 0.92, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.21, 95% CI 2-sided [-4.48 to 4.05]
Statistical Analysis 2: Comparison: Distress Screening vs No Screening; The data below is for FACT-B 6 month Total Score; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.57, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 1.37, 95% CI 2-sided [-3.41 to 6.15]
Statistical Analysis 3: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 12 month Total Score; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.62, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 1.18, 95% CI 2-sided [-3.54 to 5.89]
Statistical Analysis 4: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 3 month Physical Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.83, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.12, 95% CI 2-sided [-0.99 to 1.23]
Statistical Analysis 5: Comparison: Distress Screening vs No Screening; Data below is for the Fact-B 6 month Physical Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.82, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.15, 95% CI 2-sided [-1.15 to 1.45]
Statistical Analysis 6: Comparison: Distress Screening vs No Screening; Data below is for the Fact-B 12 month Physical Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.84, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.13, 95% CI 2-sided [-1.41 to 1.15]
Statistical Analysis 7: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 3 month Social/Family Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.77, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.17, 95% CI 2-sided [-1.31 to 0.96]
Statistical Analysis 8: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 6 month Social/Family Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.42, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.56, 95% CI 2-sided [-1.91 to 0.79]
Statistical Analysis 9: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 12 month Social/Family Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.90, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.08, 95% CI 2-sided [-1.41 to 1.24]
Statistical Analysis 10: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 3 month Emotional Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.90, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.05, 95% CI 2-sided [-0.76 to 0.87]
Statistical Analysis 11: Comparison: Distress Screening vs No Screening; The data below is for the Fact B 6 month Emotional Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.25, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.58, 95% CI 2-sided [-0.40 to 1.56]
Statistical Analysis 12: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 12 month Emotional Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.22, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.60, 95% CI 2-sided [-0.36 to 1.57]
Statistical Analysis 13: Comparison: Distress Screening vs No Screening; The data below is for Fact-B 3 month Functional Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.81, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.14, 95% CI 2-sided [-1.05 to 1.34]
Statistical Analysis 14: Comparison: Distress Screening vs No Screening; The data below is for Fact-B 6 month Functional Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.45, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.54, 95% CI 2-sided [-0.85 to 1.94]
Statistical Analysis 15: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 12 month Functional Well-Being Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.87, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.11, 95% CI 2-sided [-1.48 to 1.26]
Statistical Analysis 16: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 3 month Breast Cancer Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.80, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.16, 95% CI 2-sided [-1.13 to 1.45]
Statistical Analysis 17: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 6 month Breast Cancer Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.35, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.73, 95% CI 2-sided [-0.79 to 2.24]
Statistical Analysis 18: Comparison: Distress Screening vs No Screening; The data below is for the Fact-B 12 month Breast Cancer Subscale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.42, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.60, 95% CI 2-sided [-0.88 to 2.09]

4. Secondary Outcome: Breast Cancer Prevention Trial (BCPT) Symptom Checklist
Description: Self-reported measure of physical symptoms in the past 4 weeks; scale: 0=not at all; 1=slightly; 2=moderately; 3=quite a bit; 4=extremely. Higher scores indicate greater symptom burden. Sub-scales include Hot Flashes, Nausea, Bladder Control, Vaginal Problems, Musculoskelatal Pain, Cognitive Problems, Weight Problems, and Arm Problems.
Time Frame: 12 months
Population: Number of participants analyzed varies across rows for 3-, 6- and 12-month surveys because not all patients completed all surveys and/or answered all questions in a survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Distress Screening | No Screening
Number analyzed (Participants) | 221 | 235
units on a scale
  BCPT Survey 3 Month Total Score | 0.9 (0.6) | 1.0 (0.7)
  BCPT Survey 3 month Hot Flashes Sub-Scale: number analyzed (Participants) | 217 | 230
  BCPT Survey 3 month Hot Flashes Sub-Scale | 1.2 (1.1) | 1.2 (1.2)
  BCPT Survey 3 month Nausea Sub-Scale: number analyzed (Participants) | 216 | 231
  BCPT Survey 3 month Nausea Sub-Scale | 0.4 (0.7) | 0.5 (0.8)
  BCPT Suvey 3 month Bladder Control Sub-Scale: number analyzed (Participants) | 219 | 233
  BCPT Suvey 3 month Bladder Control Sub-Scale | 0.6 (0.9) | 0.7 (1.0)
  BCPT Survey 3 month Vaginal/Sex Problems Sub-Scale: number analyzed (Participants) | 175 | 188
  BCPT Survey 3 month Vaginal/Sex Problems Sub-Scale | 0.6 (1.0) | 0.8 (1.1)
  BCPT Survey 3 month Musculoskeletal Pain Sub-Scale: number analyzed (Participants) | 220 | 234
  BCPT Survey 3 month Musculoskeletal Pain Sub-Scale | 1.5 (1.1) | 1.5 (1.1)
  BCPT Suvey 3 month Cognitive Problems Sub-Scale: number analyzed (Participants) | 221 | 233
  BCPT Suvey 3 month Cognitive Problems Sub-Scale | 1.2 (1.0) | 1.2 (1.1)
  BCPT Survey 3 month Weight Problems Sub-Scale: number analyzed (Participants) | 212 | 231
  BCPT Survey 3 month Weight Problems Sub-Scale | 1.1 (1.0) | 1.2 (1.2)
  BCPT Survey 3 month Arm Problems Sub-Scale: number analyzed (Participants) | 213 | 227
  BCPT Survey 3 month Arm Problems Sub-Scale | 0.6 (0.8) | 0.5 (0.9)
  BCPT Suvey 6 month Total Score: number analyzed (Participants) | 123 | 127
  BCPT Suvey 6 month Total Score | 0.9 (0.7) | 0.9 (0.6)
  BCPT Survey 6 month Hot Flashes Sub-Scale: number analyzed (Participants) | 122 | 126
  BCPT Survey 6 month Hot Flashes Sub-Scale | 1.2 (1.1) | 1.1 (1.2)
  BCPT Survey 6 month Nausea Sub-Scale: number analyzed (Participants) | 122 | 126
  BCPT Survey 6 month Nausea Sub-Scale | 0.2 (0.4) | 0.3 (0.5)
  BCPT Survey 6 month Bladder Control Sub-Scale: number analyzed (Participants) | 121 | 126
  BCPT Survey 6 month Bladder Control Sub-Scale | 0.7 (1.0) | 0.6 (0.9)
  BCPT Survey 6 month Vaginal/Sex Problems Sub-Scale: number analyzed (Participants) | 94 | 103
  BCPT Survey 6 month Vaginal/Sex Problems Sub-Scale | 0.7 (1.0) | 0.8 (1.1)
  BCPT Survey 6 month Musculoskeletal Pain Sub-Scale: number analyzed (Participants) | 121 | 126
  BCPT Survey 6 month Musculoskeletal Pain Sub-Scale | 1.5 (1.1) | 1.4 (1.2)
  BCPT Survey 6 month Cognitive Problems Sub-Scale: number analyzed (Participants) | 122 | 127
  BCPT Survey 6 month Cognitive Problems Sub-Scale | 1.0 (1.0) | 1.0 (1.0)
  BCPT Survey 6 month Weight Problems Sub-Scale: number analyzed (Participants) | 120 | 125
  BCPT Survey 6 month Weight Problems Sub-Scale | 1.1 (1.1) | 1.2 (1.1)
  BCPT Survey 6 month Arm Problems Sub-Scale: number analyzed (Participants) | 114 | 121
  BCPT Survey 6 month Arm Problems Sub-Scale | 0.5 (0.7) | 0.5 (0.8)
  BCPT Survey 12 month Total Score: number analyzed (Participants) | 131 | 136
  BCPT Survey 12 month Total Score | 0.9 (0.6) | 0.9 (0.6)
  BCPT Survey 12 month Hot Flashes Sub-Scale: number analyzed (Participants) | 131 | 133
  BCPT Survey 12 month Hot Flashes Sub-Scale | 1.1 (1.1) | 1.0 (1.1)
  BCPT Survey 12 month Nausea Sub-Scale: number analyzed (Participants) | 131 | 134
  BCPT Survey 12 month Nausea Sub-Scale | 0.2 (0.4) | 0.3 (0.6)
  BCPT Survey 12 month Bladder Control Sub-Scale: number analyzed (Participants) | 131 | 133
  BCPT Survey 12 month Bladder Control Sub-Scale | 0.7 (0.9) | 0.7 (0.9)
  BCPT Survey 12 month Vaginal/Sex Problem Sub-Scale: number analyzed (Participants) | 114 | 110
  BCPT Survey 12 month Vaginal/Sex Problem Sub-Scale | 0.8 (1.1) | 0.9 (1.2)
  BCPT Survey 12 month Musculoskeletal Pain Sub-Scal: number analyzed (Participants) | 131 | 135
  BCPT Survey 12 month Musculoskeletal Pain Sub-Scal | 1.7 (1.1) | 1.5 (1.1)
  BCPT Survey 12 month Cognitive Problems Sub-Scale: number analyzed (Participants) | 131 | 136
  BCPT Survey 12 month Cognitive Problems Sub-Scale | 1.0 (1.0) | 1.1 (1.0)
  BCPT Survey 12 month Weight Problems Sub-Scale: number analyzed (Participants) | 127 | 133
  BCPT Survey 12 month Weight Problems Sub-Scale | 1.0 (1.1) | 1.1 (1.0)
  BCPT Survey 12 month Arm Problems Sub-Scale: number analyzed (Participants) | 130 | 135
  BCPT Survey 12 month Arm Problems Sub-Scale | 0.5 (0.8) | 0.5 (0.7)
Statistical Analysis 1: Comparison: Distress Screening vs No Screening; Data below is for the BCPT survey 3 month Total Score; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.59, Mixed Models Analysis — We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.03, 95% CI 2-sided [-0.15 to 0.09]
Statistical Analysis 2: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 6 month Total Score; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.47, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.05, 95% CI 2-sided [-0.09 to 0.19]
Statistical Analysis 3: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 12 month Total Score; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.37, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.06, 95% CI 2-sided [-0.20 to 0.07]
Statistical Analysis 4: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 3 month Hot Flashes Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.65, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.05, 95% CI 2-sided [-0.26 to 0.17]
Statistical Analysis 5: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 6 month Hot Flashes Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.54, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.08, 95% CI 2-sided [-0.17 to 0.33]
Statistical Analysis 6: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 12 month Hot Flashes Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.87, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.02, 95% CI 2-sided [-0.27 to 0.22]
Statistical Analysis 7: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 3 month Nausea Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.32, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.06, 95% CI 2-sided [-0.17 to 0.06]
Statistical Analysis 8: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 6 month Nausea Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.96, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.00, 95% CI 2-sided [-0.15 to 0.14]
Statistical Analysis 9: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 12 month Nausea Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.32, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.07, 95% CI 2-sided [-0.21 to 0.07]
Statistical Analysis 10: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 3 month Bladder Control Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.44, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.07, 95% CI 2-sided [-0.24 to 0.11]
Statistical Analysis 11: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 6 month Bladder Control Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.38, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.09, 95% CI 2-sided [-0.11 to 0.30]
Statistical Analysis 12: Comparison: Distress Screening vs No Screening; The data below is for the BCPT survey 12 month Bladder Control Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.47, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.07, 95% CI 2-sided [-0.28 to 0.13]
Statistical Analysis 13: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 3 month Vaginal Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.13, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.17, 95% CI 2-sided [-0.39 to 0.05]
Statistical Analysis 14: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 6 month Vaginal Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.03, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.29, 95% CI 2-sided [-0.55 to -0.02]
Statistical Analysis 15: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 12 month Vaginal Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.14, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.19, 95% CI 2-sided [-0.45 to 0.06]
Statistical Analysis 16: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 3 month Musculoskeletal Pain Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.53, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.07, 95% CI 2-sided [-0.14 to 0.28]
Statistical Analysis 17: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 6 month Musculoskeletal Pain Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.47, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.10, 95% CI 2-sided [-0.16 to 0.35]
Statistical Analysis 18: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 12 month Musculoskeletal Pain Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.57, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.07, 95% CI 2-sided [-0.18 to 0.33]
Statistical Analysis 19: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 3 month Cognitive Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.85, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.02, 95% CI 2-sided [-0.18 to 0.21]
Statistical Analysis 20: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 6 month Cognitive Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.38, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.10, 95% CI 2-sided [-0.12 to 0.32]
Statistical Analysis 21: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 12 month Cognitive Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.23, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.13, 95% CI 2-sided [-0.35 to 0.09]
Statistical Analysis 22: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 3 month Weight Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.18, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.14, 95% CI 2-sided [-0.35 to 0.07]
Statistical Analysis 23: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 6 month Weight Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.35, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.12, 95% CI 2-sided [-0.36 to 0.13]
Statistical Analysis 24: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 12 month Weight Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.34, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = -0.12, 95% CI 2-sided [-0.36 to 0.12]
Statistical Analysis 25: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 3 month Arm Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.22, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.09, 95% CI 2-sided [-0.06 to 0.25]
Statistical Analysis 26: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 6 month Arm Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.26, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.11, 95% CI 2-sided [-0.08 to 0.29]
Statistical Analysis 27: Comparison: Distress Screening vs No Screening; The data below is the BCPT survey 12 month Arm Problems Sub-Scale; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.34, Mixed Models Analysis; We used a difference-in-differences model to estimate the time, treatment, and time-by-treatment effects; see above = 0.09, 95% CI 2-sided [-0.09 to 0.27]

5. Secondary Outcome: Number of Patients With Oncology Visit
Description: Between group comparison of number of visits to oncology. Restricted to patients with at least 100 days of follow-up. Covariates included in multivariable models were age, Charlson's comorbidity index, race/ethnicity, marital status, and cancer stage.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Screening | No Screening
Number analyzed (Participants) | 730 | 683
Participants | 728 | 683
Statistical Analysis 1: Comparison: Distress Screening vs No Screening; Test type: Other; p = 0.006, Regression, Poisson; Rate Ratio = 0.86, 95% CI 2-sided [0.77 to 0.96]

6. Secondary Outcome: Number of Patients With Primary Care Visit
Description: Between group comparison of number of visits to primary care. Restricted to patients with at least 100 days of follow-up. Covariates included in multivariable models were age, Charlson's comorbidity index, race/ethnicity, marital status, and cancer stage.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Screening | No Screening
Number analyzed (Participants) | 730 | 683
Participants | 648 | 616
Statistical Analysis 1: Comparison: Distress Screening vs No Screening; Test type: Other; p = 0.356, Regression, Poisson; Rate Ratio = 1.07, 95% CI 2-sided [0.93 to 1.07]

7. Other Pre Specified Outcome: Number of Participants Utilizing Behavioral Health Services
Description: Between group comparison of number of visits with behavioral health providers. Restricted to patients with at least 100 days of follow-up. Covariates included in multivariable models were age, Charlson's comorbidity index, race/ethnicity, marital status, and cancer stage.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Screening | No Screening
Number analyzed (Participants) | 730 | 683
Participants | 287 | 247
Statistical Analysis 1: Comparison: Distress Screening vs No Screening; Test type: Other; p = 0.919, Regression/Poisson; Rate Ratio = 1.02, 95% CI 2-sided [0.73 to 1.41]

8. Other Pre Specified Outcome: Number of Participants Utilizing Emergency and Urgent Care Services
Description: Between group comparison of number of visits to emergency and urgent care services. Restricted to patients with at least 100 days of follow-up. Covariates included in multivariable models were age, Charlson's comorbidity index, race/ethnicity, marital status, and cancer stage.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Distress Screening | No Screening
Number analyzed (Participants) | 730 | 683
Participants
  ED Visits | 248 | 213
  Urgent Care Visits | 269 | 279
Statistical Analysis 1: Comparison: Distress Screening vs No Screening; The data below applies to Emergency Department visits; Test type: Other; p = 0.367, Regression, Poisson; Rate Ratio = 1.16, 95% CI 2-sided [0.84 to 1.62]
Statistical Analysis 2: Comparison: Distress Screening vs No Screening; The data below applies to Urgent Care visits; Test type: Other; p = 0.497, Regression, Poisson; Rate Ratio = 0.84, 95% CI 2-sided [0.51 to 1.38]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Distress Screening | No Screening
All-Cause Mortality (participants affected / at risk) | 25/744 | 16/692
Serious Adverse Events (participants affected / at risk) | 0/744 | 0/692
Other Adverse Events (participants affected / at risk) | 0/744 | 0/692

LIMITATIONS AND CAVEATS:
No limitations to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT02941614/Prot_SAP_000.pdf